CLINICAL TRIAL: NCT03221257
Title: Scleroderma Lung Study III (SLS III): Combining the Anti-fibrotic Effects of Pirfenidone (PFD) With Mycophenolate (MMF) for Treating Scleroderma-related Interstitial Lung Disease
Brief Title: Scleroderma Lung Study III - Combining Pirfenidone With Mycophenolate
Acronym: SLSIII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Roth (Other)
Collaborators: University of Michigan (Other); Genentech, Inc. (Industry); University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Michael Roth, Professor of Pulmonary and Critical Care Medicine, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCLA-SLS3
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Scleroderma, Systemic; Interstitial Lung Disease
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial | interventions — pirfenidone; 5'-palmitoyl cytarabine; Mycophenolic Acid; Drugs, Generic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Plac) + Mycophenolate (MMF) (Placebo Comparator): Participants will receive Placebo (Plac) as add-on to a background therapy of Mycophenolate Mofetil (MMF).
  Interventions: Drug: Placebo (Plac); Drug: Mycophenolate Mofetil (MMF)
- Pirfenidone (PFD) + Mycophenolate (MMF) (Experimental): Participants will receive Pirfenidone (PFD) as add-on to a background therapy of Mycophenolate Mofetil (MMF).
  Interventions: Drug: Pirfenidone (PFD); Drug: Mycophenolate Mofetil (MMF)

INTERVENTIONS:
Drug: Pirfenidone (PFD) — Participants will receive PFD titrated up to a target dose of 801 mg taken three times daily as tolerated (3-step titration occurring at 2 week intervals).
  Other Names: Esbriet
  Arms: Pirfenidone (PFD) + Mycophenolate (MMF)
Drug: Placebo (Plac) — Participants will receive a Plac, matched to resemble PFD, titrated up to a target dose of 801 mg taken three times daily as tolerated (3-step titration occurring at 2 week intervals).
  Other Names: Inactive capsule
  Arms: Placebo (Plac) + Mycophenolate (MMF)
Drug: Mycophenolate Mofetil (MMF) — Participants will receive MMF titrated up to a target dose of 1500 mg taken twice daily as tolerated (4-step titration occurring at monthly intervals).
  Other Names: generic for Cellcept

SUMMARY:
A Phase II multi-center, double-blind, parallel group, randomized and placebo-controlled clinical trial addressing the treatment of patients with active and symptomatic Scleroderma-related interstitial lung disease (SSc-ILD).

DETAILED DESCRIPTION:
A Phase II multi-center, double-blind, parallel group, randomized and placebo-controlled clinical trial addressing the treatment of patients with active and symptomatic Scleroderma-related interstitial lung disease (SSc-ILD). Patients who are either treatment naive or only recently started treatment (</= 6 months of prior treatment) will be randomized in a 1:1 assignment to receive either oral mycophenolate mofetil (MMF) and a placebo (Plac) or a combination of oral MMF and oral pirfenidone (PFD), with both regimens administered for 18 months. The primary hypothesis is that the rapid onset and anti-fibrotic effects of PFD, which have been observed in the treatment of Idiopathic Pulmonary Fibrosis (IPF), will complement the delayed antiinflammatory and immunosuppressive effects of MMF, to produce a significantly more rapid and/or greater improvement in lung function over time than occurs in patients receiving control therapy with MMF and Plac.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 yrs
2. Scleroderma as determined by the 2013 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria.
3. Grade ≥2 on the Magnitude of Task component of the Mahler Modified Dyspnea Index
4. FVC-% of ≤85% at screening
5. Onset of the first non-Raynaud manifestation of SSc within the prior 84 months.
6. Presence of any ground-glass opacification (GGO) on thoracic high-resolution computed tomography (HRCT)
7. Repeat FVC-% at the baseline visit within 10% of the FVC-% value measured at screening. If these criteria are not met, a repeat FVC-% may be obtained within 7 days and the subject may qualify for randomization if the repeat FVC-% agrees within 10% of the FVC-% obtained at screening.

Exclusion Criteria:

1. Disease features supporting the primary diagnosis of another connective tissue disease such as rheumatoid arthritis, systemic lupus erythematosus or mixed connective tissue disease (Features consistent with a secondary Sjogren syndrome or scleroderma-associated myopathy will be allowed).
2. FVC-% of <45% at either screening or baseline.
3. Forced Expiratory Volume in the first second (FEV1)/Forced Vital Capacity (FVC) ratio <0.65 at either screening or baseline.
4. Diffusing capacity of the lung for carbon monoxide adjusted for hemoglobin, expressed as a percentage of the normal predicted value (DLCOHb-%) of <30% at screening or <25% at baseline.

   a) All participants with a DLCOHb-% between 30 to 40% must have pulmonary artery pressures documented by either echocardiogram, right heart catheterization or magnetic resonance imaging in order to be considered for inclusion.
5. Diagnosis of clinically significant resting pulmonary hypertension requiring treatment or mild pulmonary hypertension requiring treatment with more than one oral medication as ascertained prior to study evaluation or as part of a standard of care clinical assessment performed outside of the study protocol.
6. Evidence of uncontrolled congestive heart failure, unstable ischemic heart disease, history of complicated pulmonary embolism impacting on heart or lung function, or unstable cardiac arrhythmia requiring chronic anticoagulation.
7. Clinically significant abnormalities on HRCT not attributable to SSc
8. Hematologic abnormality at screening including:

   1. Leukopenia (white blood cells [WBC] <4.0x10^3/µl).
   2. Thrombocytopenia (platelet count <120.0x10^3/µl).
   3. Clinically significant anemia [Hemoglobin (Hgb) <10.0 g/dl].

   Participants with an identified and correctable etiology may be eligible if repeat testing within the maximal 90-day screening period meets all criteria.
9. A diagnosis of chronic liver disease or abnormal baseline liver function test (LFTs) or total bilirubin that are >2.0 x upper normal limit
10. Serum creatinine >2.0mg/dl
11. History of recurrent aspiration, uncontrolled heartburn, or gastroesophageal reflux disease (GERD) with a reflux scale score of >1.00 as determined by a UCLA Scleroderma Clinical Trial Consortium Gastrointestinal Scale (UCLA SCTC GIT), Version 2.0.

    Participants with uncontrolled heartburn or GERD that is amenable to medical management may be eligible if repeat testing within the maximal 90-day screening period meets this criteria.
12. Known achalasia, esophageal stricture or esophageal dysfunction sufficient to limit the ability to swallow medication.
13. Pregnancy (as documented by blood test) and/or breast feeding
14. If of child bearing potential (a female participant < 55 years of age who has not been postmenopausal for ≥ 5 years or who has not had a bilateral salpingectomy, hysterectomy and/or oophorectomy), failure to employ two reliable means of contraception which may include surgical sterilization, barrier methods, spermicides, intrauterine devices, and/or hormonal contraception, unless the participant chooses abstinence (to avoid heterosexual intercourse completely). If a subject chooses abstinence, then a second reliable means of contraception is not needed.
15. Prior use of potential disease modifying antirheumatic drugs (DMARDs) according to the following exposure rules:

    1. Use of oral cyclophosphamide (CYC), MMF, azathioprine or other oral or short half-life DMARDs (as detailed in Protocol Section 7.5.1a) for more than 6 months in the past year as determined at the time of the initial screening visit.
    2. Treatment with more than three intravenous doses of CYC, one treatment course of Rituximab or other intravenous or injectable DMARDs (as detailed in Protocol Section 7.5.1b) in the past year.
    3. More distant history of treatment with a DMARD is allowed as long as the patient has a new diagnosis/new episode of active SSc-ILD since stopping that treatment and meets the criteria noted in 15a or 15b.
16. Use of CYC, MMF, azathioprine, Rituximab or other DMARD (as defined in Protocol Section 7.5.1a&b) in the 30 days prior to their baseline visit unless the patient is on MMF and the responsible physician indicates that continued use is in the best clinical interest of the patient.
17. Active infection (lung, ulcers or elsewhere) whose management would be compromised by immunosuppression.
18. Other serious concomitant medical illness (e.g., active malignancy within the past 5 years other than surgically-removed local skin cancer such as a basal cell carcinoma), chronic debilitating illness (other than SSc), unreliability or drug abuse that might compromise the patient's participation in the trial.
19. Current use, or use within the 30 days prior to their baseline visit, of prednisone (or equivalent) in doses >10 mg/day.
20. Smoking of cigars, pipes, or cigarettes during the past 6 months.
21. Use of contraindicated medications, including medications with putative disease-modifying properties that do not meet the exposure limits described in Exclusion Criteria #15 and #16, moderate or strong inhibitors of cytochrome P450 (CYP) isozyme 1A2 (CYP1A2) (note ciprofloxacin allowed up to a dose of 500 mg twice daily), and moderate inducers of CYP1A2 (such as tobacco smoke or phenytoin). See Protocol Section 7.5 for complete list.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Roth, MD, Principal Investigator — Pulmonary & Critical Care Medicine, Geffen School of Medicine at UCLA
Locations (16):
- United States (16):
  - University of California Los Angeles, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard Medical School, Brigham & Women's Hospital, Boston, Massachusetts
  - Boston University, School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Rutgers University, New Brunswick, New Jersey
  - Hospital for Special Surgery, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Medical School at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
A bio-specimen repository will be created in which de-identified blood specimens will be made available to qualified researchers who submit meritorious applications for the access and use of such samples. Requests for specimens and correlative analyses related to other linked and de-identified clinical data will be overseen by the Study Executive and Steering Committees and/or any sub-committees that they may appoint for this process.
Time Frame: Sharing will be made available after completion of the clinical trial and reporting of the primary outcome.
Access Criteria: Access criteria will be made available after 01/01/2018 through the study website noted below.
URL: http://sclerodermalungstudy.org

REFERENCES:
- [Background] Tashkin DP, Roth MD, Clements PJ, Furst DE, Khanna D, Kleerup EC, Goldin J, Arriola E, Volkmann ER, Kafaja S, Silver R, Steen V, Strange C, Wise R, Wigley F, Mayes M, Riley DJ, Hussain S, Assassi S, Hsu VM, Patel B, Phillips K, Martinez F, Golden J, Connolly MK, Varga J, Dematte J, Hinchcliff ME, Fischer A, Swigris J, Meehan R, Theodore A, Simms R, Volkov S, Schraufnagel DE, Scholand MB, Frech T, Molitor JA, Highland K, Read CA, Fritzler MJ, Kim GHJ, Tseng CH, Elashoff RM; Sclerodema Lung Study II Investigators. Mycophenolate mofetil versus oral cyclophosphamide in scleroderma-related interstitial lung disease (SLS II): a randomised controlled, double-blind, parallel group trial. Lancet Respir Med. 2016 Sep;4(9):708-719. doi: 10.1016/S2213-2600(16)30152-7. Epub 2016 Jul 25. PMID 27469583
- [Background] Tashkin DP, Volkmann ER, Tseng CH, Roth MD, Khanna D, Furst DE, Clements PJ, Theodore A, Kafaja S, Kim GH, Goldin J, Ariolla E, Elashoff RM. Improved Cough and Cough-Specific Quality of Life in Patients Treated for Scleroderma-Related Interstitial Lung Disease: Results of Scleroderma Lung Study II. Chest. 2017 Apr;151(4):813-820. doi: 10.1016/j.chest.2016.11.052. Epub 2016 Dec 22. PMID 28012804
- [Background] Volkmann ER, Tashkin DP, Li N, Roth MD, Khanna D, Hoffmann-Vold AM, Kim G, Goldin J, Clements PJ, Furst DE, Elashoff RM. Mycophenolate Mofetil Versus Placebo for Systemic Sclerosis-Related Interstitial Lung Disease: An Analysis of Scleroderma Lung Studies I and II. Arthritis Rheumatol. 2017 Jul;69(7):1451-1460. doi: 10.1002/art.40114. Epub 2017 May 23. PMID 28376288
- [Background] Namas R, Tashkin DP, Furst DE, Wilhalme H, Tseng CH, Roth MD, Kafaja S, Volkmann E, Clements PJ, Khanna D; Participants in the Scleroderma Lung Study I and members of the Scleroderma Lung Study II Research Group. Efficacy of Mycophenolate Mofetil and Oral Cyclophosphamide on Skin Thickness: Post Hoc Analyses From Two Randomized Placebo-Controlled Trials. Arthritis Care Res (Hoboken). 2018 Mar;70(3):439-444. doi: 10.1002/acr.23282. Epub 2018 Feb 9. PMID 28544580
- [Background] Khanna D, Albera C, Fischer A, Khalidi N, Raghu G, Chung L, Chen D, Schiopu E, Tagliaferri M, Seibold JR, Gorina E. An Open-label, Phase II Study of the Safety and Tolerability of Pirfenidone in Patients with Scleroderma-associated Interstitial Lung Disease: the LOTUSS Trial. J Rheumatol. 2016 Sep;43(9):1672-9. doi: 10.3899/jrheum.151322. Epub 2016 Jul 1. PMID 27370878
- [Background] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312
- [Derived] Takizawa A, Kamita M, Kondoh Y, Bando M, Kuwana M, Inoue Y. Current monitoring and treatment of progressive fibrosing interstitial lung disease: a survey of physicians in Japan, the United States, and the European Union. Curr Med Res Opin. 2021 Feb;37(2):327-339. doi: 10.1080/03007995.2020.1860920. Epub 2021 Jan 11. PMID 33287583

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 88 consented with 31 subsequently deemed ineligible, 6 withdrawals prior to randomization, resulting in 51 participants considered enrolled, eligible and randomized.
Period: Overall Study
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Started | 24 | 27
Completed | 23 | 25
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population includes all the randomized participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF) | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (10) | 56.6 (9.9) | 54.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 19 | 22 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51
Scleroderma Classification [Count of Participants; unit: Participants]
  Sine | 3 | 3 | 6
  Limited | 13 | 11 | 24
  Diffuse | 8 | 13 | 21
Disease Duration [Mean (Standard Deviation); unit: months] — Population: The disease duration was not available for all participants.
  months
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 32.9 (24.2) | 28.9 (25.4) | 30.8 (24.7)
Percent predicted forced vital capacity (FVC-%) [Mean (Standard Deviation); unit: percent predicted] | 71.5 (9.9) | 70.6 (11.0) | 71.0 (10.4)
Forced Vital Capacity volume (FVC) [Mean (Standard Deviation); unit: ml] | 2705 (540) | 2610 (781) | 2655 (674)
Percent predicted single-breath diffusing capacity for carbon monoxide (DLCOHb-%) [Mean (Standard Deviation); unit: percent predicted] — Population: DLCOHb-% was not available for all participants.
  percent predicted
    number analyzed (Participants) | 24 | 26 | 50
    (all) | 55.6 (14.4) | 54.6 (12.0) | 55.1 (13.0)
Mahler Baseline Dyspnea Index [Mean (Standard Deviation); unit: units on a scale] — Mahler Baseline Dyspnea Index (BDI) measures the level of dyspnea at baseline, ranging from 0 to 12. The lower the score indicates the greater severity of dyspnea.
  units on a scale | 6.8 (1.5) | 6.9 (2.0) | 6.9 (1.8)
Modified Rodnan Skin Score (mRSS) [Mean (Standard Deviation); unit: units on a scale] — The modified Rodnan Skin Score (mRSS) assesses skin thickness at each of 17 body areas, with each site scored from 0-3 (0 = normal; 1= mild thickness; 2 = moderate; 3 = severe thickness). The composite score ranges from 0 to 51, with a higher score indicating more severe skin involvement.
  units on a scale | 8.1 (7.6) | 11.7 (9.9) | 10.0 (9.0)
Health Assessment Questionnaire Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire-Disability Index (HAQ-DI) is a self-reported questionnaire covering eight domains related to difficulty in performing activities of daily living. The index score ranges 0-3, with a higher number indicating worse disability.
  units on a scale | 0.4 (0.4) | 0.5 (0.6) | 0.5 (0.5)
Quantitative lung fibrosis score in the whole lung (QLF-WL) [Mean (Standard Deviation); unit: percent] — The Quantitative Lung Fibrosis Score in the Whole Lung (QLF-WL) represents the percentage of imaging pixels within the whole lung (WL), obtained from a volumetric high resolution computerized tomography (HRCT) scan and scored by a computer algorithm, that exhibit features characteristic for lung fibrosis. Score ranges 0 to 100% with higher percentages representing greater extent of lung fibrosis. Population: HRCT data was not available for all participants.
  percent
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 6.0 (5.1) | 6.5 (6.0) | 6.3 (5.5)
Quantitative lung fibrosis score in the lobe of maximal involvement (QLF-LM) [Mean (Standard Deviation); unit: percent] — Lobes on HRCT images are analyzed using a computer algorithm to determine the percentage of overall pixels exhibiting features characteristic for quantitative lung fibrosis (QLF). Quantitative Lung Fibrosis in the Lobe of Maximal Involvement (QLF-LM) is the maximum score among the lobes, indicating the most severe lobe. Score ranges 0 to 100% with higher percentages representing greater involvement of QLF. Population: HRCT data was not available for all participants.
  percent
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 14.5 (14.0) | 16.3 (17.4) | 15.4 (15.7)
Quantitative interstitial lung disease score in the whole lung (QILD-WL) [Mean (Standard Deviation); unit: percent] — The Quantitative Interstitial Lung Disease Score in the Whole Lung (QILD-WL) represents the percentage of imaging pixels within the WL, obtained from a volumetric HRCT scan, that exhibit features of any three patterns of interstitial lung disease (ILD) including quantitative ground-glass opacity (QGG), lung fibrosis (QLF) and quantitative honeycombing (QHC). Score ranges 0 to 100% with higher percentages representing greater extent of ILD. Population: HRCT data was not available for all participants.
  percent
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 24.1 (11.3) | 23.8 (11.8) | 23.9 (11.4)
Quantitative interstitial lung disease score in the lobe of maximal involvement (QILD-LM) [Mean (Standard Deviation); unit: percent] — Lobes on HRCT images are analyzed using a computer algorithm to determine the percentage of overall pixels exhibiting features characteristic for any of three patterns of ILD including QGG, QLF and QHC. Quantitative Interstitial Lung Disease in the Lobe of Maximal Involvement (QILD-LM) is the maximum score among the lobes, indicating the most severe lobe. Score ranges 0 to 100% with higher percentages representing greater extent of ILD. Population: HRCT data was not available for all participants.
  percent
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 42.0 (17.9) | 41.8 (19.5) | 41.9 (18.6)
Total lung capacity (TLC) [Mean (Standard Deviation); unit: ml] — Total Lung Capacity (TLC) is the volume of air in the lungs, determined by computer-aided measurement of lung volume on a volumetric HRCT performed at maximal inspiratory breath hold. Score represents a continuous value, in milliliters, with the higher number indicating greater volume. Population: HRCT data was not available for all participants.
  ml
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 3859 (883) | 3717 (874) | 3783 (872)

OUTCOME MEASURES:

1. Primary Outcome: Percent Predicted Forced Vital Capacity (FVC-%)
Description: Change from baseline to month 18 in the mean forced vital capacity (represented as the percentage of the age-; height-; gender-; and race-adjusted predicted value, i.e. FVC-%).
Time Frame: Baseline to 18 months
Population: The modified intention-to-treat population (m-ITT) is defined as all participants randomized, receiving at least one dose of study medication, and having at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: percent predicted
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 24 | 27
percent predicted | 2.24 (1.351) | 2.09 (1.278)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.9326, Mixed Models Analysis; Mean Difference (Net) = -0.14

2. Other Pre Specified Outcome: Percent Predicted Single-breath Diffusing Capacity for Carbon Monoxide (DLCOHb-%)
Description: Change from baseline to month 18 in DLCO, calculated as a percent of the age-; height-; gender-; race-; and hemoglobin-adjusted predicted value (DLCOHb-%). The raw DLCO value and adjusting it for all of these factors and presenting it as a percent of predicted (expected) is the outcome measure (DLCOHb-%).
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent predicted
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 24 | 25
percent predicted | 1.25 (1.549) | 1.24 (1.505)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.9968, Mixed Models Analysis; Mean Difference (Net) = -0.01

3. Other Pre Specified Outcome: Modified Rodnan Skin Score (mRSS)
Description: Change from baseline to month 18 in the mRSS. mRSS scores have a range from 0 to 51, with higher score indicating greater skin involvement.
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 24 | 27
score on a scale | -5.42 (1.164) | -4.96 (1.109)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.7489, Mixed Models Analysis; Mean Difference (Net) = 0.46

4. Other Pre Specified Outcome: Forced Vital Capacity Volume (FVC, in ml)
Description: Change from baseline to month 18 in the Forced Vital Capacity volume (FVC, in ml)
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ml
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 24 | 27
ml | 121.53 (62.41) | 112.33 (59.055)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.8898, Mixed Models Analysis; Mean Difference (Net) = -9.2

5. Other Pre Specified Outcome: Mahler Modified Transitional Dyspnea Index (TDI)
Description: The change from baseline to 18 months in dyspnea. The TDI score for each of three domains ranges from -3 (major deterioration) to +3 (major improvement). The sum of all domains yields the TDI total score (-9 to +9).
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 24 | 27
score on a scale | 1.13 (0.754) | 1.99 (0.710)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.3826, Mixed Models Analysis; Mean Difference (Net) = 0.86

6. Other Pre Specified Outcome: Health Assessment Questionnaire Modified for Scleroderma (HAQ-DI)
Description: Change from baseline to month 18 as a subjective measure of dyspnea and quality of life.
  HAQ-DI ranges from 0 (no disability) to 3 (severe disability).
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 23 | 26
score on a scale | -0.03 (0.109) | -0.17 (0.103)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.2819, Mixed Models Analysis; Mean Difference (Net) = -0.14

7. Other Pre Specified Outcome: St. George's Respiratory Questionnaire (SGRQ)
Description: Change from baseline to month 18 as a subjective measure of dyspnea and quality of life. SGRQ ranges from 0 (no impairment) to 100 (maximum impairment).
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 24 | 27
score on a scale | -4.77 (3.487) | -6.11 (3.212)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.7534, Mixed Models Analysis; Mean Difference (Net) = -1.35

8. Other Pre Specified Outcome: High Resolution Computerized Tomography (HRCT) Measures of Quantitative Lung Fibrosis Score in the Whole Lung (QLF-WL)
Description: Change from screening to month 18 in computer-generated scoring of HRCT data from the whole lung for the percentage of imaging pixels that exhibit features characteristic for lung fibrosis.
  Individual image scores range 0 to 100%, with higher percentages representing greater extent of quantitative lung fibrosis.
Time Frame: Screening to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 20 | 24
percent | 1.46 (0.994) | -0.11 (0.935)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.1701, ANCOVA; Mean Difference (Net) = -1.58

9. Other Pre Specified Outcome: High Resolution Computerized Tomography (HRCT) Measures of Quantitative Lung Fibrosis Score in the Lobe of Maximal Involvement (QLF-LM)
Description: Change from screening to month 18 in computer-generated scoring of HRCT data for the percentage of imaging pixels that exhibit features characteristic for lung fibrosis within the lobe of maximal involvement at baseline.
  Individual image score range 0 to 100%, with higher percentages representing greater extent of quantitative lung fibrosis.
Time Frame: Screening to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 20 | 24
percent | 2.57 (2.276) | 0.13 (2.132)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.3515, ANCOVA; Mean Difference (Net) = -2.44

10. Other Pre Specified Outcome: High Resolution Computerized Tomography (HRCT) Measures of Quantitative Interstitial Lung Disease Score in the Whole Lung (QILD-WL)
Description: Change from screening to month 18 in computer-generated scoring of HRCT data from the whole lung for the percentage of imaging pixels that exhibit features of any of the three patterns of interstitial lung disease (ILD) including quantitative ground-glass opacity (QGG), lung fibrosis (QLF) and quantitative honeycombing (QHC).
  Individual image scores range 0 to 100%, with higher percentages representing greater extent of quantitative interstitial lung disease.
Time Frame: Screening to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 20 | 24
percent | 2.36 (1.919) | -1.15 (1.829)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.1177, ANCOVA; Mean Difference (Net) = -3.51

11. Other Pre Specified Outcome: High Resolution Computerized Tomography (HRCT) Measures of Quantitative Interstitial Lung Disease Score in the Lobe of Maximal Involvement (QILD-LM)
Description: Change from screening to month 18 in computer-generated scoring of HRCT data for the percentage of imaging pixels exhibiting features characteristic for any of three patterns of ILD (including QGG, QLF and QHC) within the lobe of maximal involvement at baseline.
  Individual image scores range 0 to 100%, with higher percentages representing greater extent of quantitative interstitial lung disease.
Time Frame: Screening to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 20 | 24
percent | 2.99 (2.634) | -0.99 (2.486)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.1931, ANCOVA; Mean Difference (Net) = -3.98

12. Other Pre Specified Outcome: High Resolution Computerized Tomography (HRCT) Measures of Total Lung Capacity (TLC)
Description: Change from screening to 18 months in quantitative HRCT measurement of TLC at maximal inspiration (HRCT-TLC).
  Higher scores indicates a better outcome.
Time Frame: Screening to 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ml
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 20 | 24
ml | 70.69 (78.986) | 191.99 (73.738)
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.1811, ANCOVA; Mean Difference (Net) = 121.30

13. Other Pre Specified Outcome: 3.0% or Greater Improvement From Baseline in FVC-%.
Description: The time (in months) required for each treatment arm to achieve a 3.0% or greater improvement from baseline in the FVC-% over the 18-month treatment period.
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 24 | 27
months | 17.8 [8.9 to NA] — Due to the fact that the number of events is insufficient to calculate the upper confidence limit. | 12.3 [3.6 to 18.3]
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.3261, Stratified log rank; Hazard Ratio (HR) = 1.433

14. Other Pre Specified Outcome: Greater Than 5% Improvement in FVC-%
Description: The percentage of subjects in each treatment arm achieving greater than a 5% improvement in FVC-% over the 18-month treatment period.
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 22 | 23
Participants | 6 | 9
Statistical Analysis 1: Comparison: Placebo (Plac) + Mycophenolate (MMF) vs Pirfenidone (PFD) + Mycophenolate (MMF); Test type: Superiority; p = 0.454, Regression, Logistic; Odds Ratio (OR) = 1.6

15. Other Pre Specified Outcome: Percentage of Participants Achieving Specified Absolute Changes of FVC-%
Description: The percentage of participants in each treatment arm achieving either improvements in the absolute change of FVC-% from baseline to 18 months by up to 5%, from 5% to <10% and from 10% to <15% or worsening by up to 5%, from 5% to <10% and from 10% to <15%.
  The descriptive analysis is presented.
Time Frame: Baseline to 18 months
Population: Completers population for FVC-% includes all subjects in the modified intent-to-treat population who had an 18-month FVC-% (regardless of completion of study medication).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 22 | 23
Participants
  ≥ 10% to < 15% | 1 | 1
  ≥ 5% to < 10% | 5 | 8
  > 0% to < 5% | 10 | 6
  > -5% to ≤ 0% | 5 | 6
  > -10% to ≤ -5% | 1 | 2

16. Other Pre Specified Outcome: Percentage of Participants Achieving Specified Absolute Changes of FVC-% Defined as Positive or Negative Responders
Description: The percentage of participants in each treatment arm who are defined as positive responders (improved at least 3% or more) or negative responders (worsened at least 3% or more), and stable (>-3% to <3%).
  The descriptive analysis is presented.
Time Frame: Baseline to 18 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 22 | 23
Participants
  Positive responder (≥ 3%) | 8 | 11
  Stable (> -3 to < 3) | 10 | 8
  Negative responder (≤ -3%) | 4 | 4

17. Other Pre Specified Outcome: Percentage of Participants Achieving Specified Absolute Changes of FVC-% Defined as Any Responders or Any Non-responders
Description: The percentage of participants in each treatment arm who are defined as any responders (improved >0%) or any non-responders (worsened </=0%).
  The descriptive analysis is presented.
Time Frame: Baseline to 18 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 22 | 23
Participants
  Responder (> 0%) | 16 | 15
  Non-responder (≤ 0%) | 6 | 8

18. Other Pre Specified Outcome: Percentage of Participants Achieving Specified Absolute Changes of mRSS
Description: The percentage of participants in each treatment arm achieving changes in 4 point increments: worsen (1 to 4, >/=5), no change (=0), improved (</=-13, -12 to -9, -8 to -5, -4 to -1).
  The descriptive analysis is presented.
Time Frame: Baseline to 18 months
Population: Completers population for mRSS includes all subjects in the modified intent-to-treat population who had an 18-month mRSS (regardless of completion of study medication).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 20 | 23
Participants
  ≤ -13 | 2 | 6
  -12 to -9 | 1 | 0
  -8 to -5 | 4 | 4
  -4 to -1 | 8 | 9
  0 | 3 | 3
  1 to 4 | 1 | 1
  ≥ 5 | 1 | 0

19. Other Pre Specified Outcome: Percentage of Participants Achieving Specified Absolute Changes of mRSS Defined as Improved, no Change and Decreased.
Description: The percentage of participants in each treatment arm achieving changes defined as improved (</=-5), no change (-5 to 5), and decreased (>5).
  The descriptive analysis is presented.
Time Frame: Baseline to 18 months
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 20 | 23
Participants
  Worsening (change > 5) | 0 | 0
  No Change (-5 ≤ change ≤ 5) | 15 | 13
  Improvement (change < -5) | 5 | 10

20. Other Pre Specified Outcome: Percentage of Participants Achieving Specified TDI Focal Score at 18 Months
Description: The percentage of participants in each treatment arm achieving either improvements in the TDI focal score at 18 months by 1-3, 4-6 and 7-9 points, no change (0) and worsened by 1-3, 4-6and 7-9 points.
  The descriptive analysis is presented.
Time Frame: 18 months
Population: Completers population for TDI includes all subjects in the modified intent-to-treat population who had an 18-month TDI (regardless of completion of study medication).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 23 | 25
Participants
  7 to 9 | 0 | 0
  4 to 6 | 1 | 1
  1 to 3 | 4 | 5
  0 | 8 | 8
  -3 to -1 | 6 | 2
  -6 to -4 | 3 | 5
  -9 to -7 | 1 | 4

21. Other Pre Specified Outcome: Percentage of Participants Achieving Specified TDI Focal Score at 18 Months Defined as Improved, no Change or Deterioration
Description: The percentage of participants in each treatment arm achieving TDI focal scores defined as improved (>0), no change and deterioration (<0).
  The descriptive analysis is presented.
Time Frame: 18 months
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 23 | 25
Participants
  Worsening (change < 0) | 5 | 6
  No Change (change = 0) | 8 | 8
  Improvement (change > 0) | 10 | 11

22. Other Pre Specified Outcome: Time to Withdrawal From the Study Drug or Treatment Failure
Description: The time from start of treatment to withdrawal or removal from active drug therapy (MMF or Plac/PFD separately) for any reason will be plotted over the course of the 18-month treatment as a measure of tolerability and toxicity. Median times to withdrawal are not available for reporting as less than half of the participants discontinued the study drugs.
Time Frame: Baseline to 18 months
Population: Safety population includes all the randomized participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 24 | 27
days | NA [NA to NA] — Insufficient number of events to calculate the median, lower, or upper confidence limit. | NA [NA to NA] — Insufficient number of events to calculate the median, lower, or upper confidence limit.

23. Other Pre Specified Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by System Organ Classification Using Preferred Medical Dictionary for Regulatory Activities (MedDRA) Terms.
Description: Adverse Events (AE) and Serious Adverse Events (SAE), classified according to preferred MedDRA terms, were systematically recorded over the course of the 18-month treatment period as a measure of toxicity. Total number of participants experiencing adverse events reported here. Complete breakdown of AE and SAE by MedDRA terms is reported in the Adverse Events section.
Time Frame: Baseline to 18 months
Population: Safety population includes all the randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
Number analyzed (Participants) | 24 | 27
Participants | 23 | 27

ADVERSE EVENTS:
Time Frame: 1 year and 6 months
Arm/Group | Placebo (Plac) + Mycophenolate (MMF) | Pirfenidone (PFD) + Mycophenolate (MMF)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/24 | 4/27
Other Adverse Events (participants affected / at risk) | 23/24 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Plac) + Mycophenolate (MMF) (N=24) | Pirfenidone (PFD) + Mycophenolate (MMF) (N=27)
Right Sided Chest Pain (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Covid-19 Infection (Infections and infestations) | 1 | 0
Herpes Zoster Ophthalmicus (Infections and infestations) | 0 | 1
Basal Cell Carcinoma, Nodular (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Extra-nodal Marginal Zone B-cell Lymphoma of the Stomach and Antrum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Scleroderma Renal Crisis (Renal and urinary disorders) | 0 | 1
Acute Chronic Hypoxemic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Plac) + Mycophenolate (MMF) (N=24) | Pirfenidone (PFD) + Mycophenolate (MMF) (N=27)
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Chest Pain (Cardiac) (Cardiac disorders) | 2 | 0
Dry Eyes (Eye disorders) | 4 | 0
Abdominal Pain (Gastrointestinal disorders) | 5 | 4
Bloating (Gastrointestinal disorders) | 1 | 3
Blood in Stool (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 10 | 12
Dysphagia (Gastrointestinal disorders) | 2 | 2
Gastro-esophageal Reflux Disease (GERD) (Gastrointestinal disorders) | 2 | 2
Heartburn (Gastrointestinal disorders) | 1 | 2
Loose Stools (Gastrointestinal disorders) | 0 | 2
Loss of Appetite (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 22
Stomach Pain (Gastrointestinal disorders) | 1 | 2
Upset Stomach (Gastrointestinal disorders) | 2 | 1
Vomiting (Emesis) (Gastrointestinal disorders) | 4 | 11
Worsening GERD (Gastrointestinal disorders) | 0 | 2
Dizziness (General disorders) | 1 | 5
Fatigue (General disorders) | 5 | 8
Fever (General disorders) | 3 | 0
Headache (General disorders) | 5 | 6
Insomnia (General disorders) | 1 | 4
ALT Increased (Hepatobiliary disorders) | 1 | 2
COVID-19 (Infections and infestations) | 0 | 4
Sinusitis (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (URI) (Infections and infestations) | 2 | 2
Urinary Tract Infection (UTI) (Infections and infestations) | 0 | 2
Yeast Infection (Infections and infestations) | 0 | 2
Weight Loss (Metabolism and nutrition disorders) | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 2
Tremors (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 3
Depression (Psychiatric disorders) | 1 | 2
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 1 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Cold (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper Respiratory Tract Infection (URI) (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Photosensitivity Reaction/Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritis (Itching) (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Only 51 (34%) of our planned recruitment goal of 150 were randomized. During the recruitment period MMF became a standard of care for treatment in early systemic sclerosis (SSc)-ILD, including the treatment of both lung and skin disease, thereby increasing the difficulty in recruiting treatment-naïve patients. Other barriers to recruitment included the Coronavirus Disease 2019 (COVID-19) epidemic and FDA approval of nintedanib as an alternative treatment during the initial phase of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03221257/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT03221257/SAP_001.pdf